CLINICAL TRIAL: NCT00372879
Title: Randomized Crossover Design Trial of Vitamin E vs Placebo for Treatment of Cramps in Amyotrophic Lateral Sclerosis.
Brief Title: Clinical Trial of Vitamin E to Treat Muscular Cramps in Patients With ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Strong, Professor Department of Clinical Neurological Sciences, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-06-451; ALSClin-001
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; vitamin E; muscle cramp
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscle Cramp | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crossover group 1 (Experimental): Vitamin E first and placebo second
  Interventions: Dietary Supplement: Vitamin E
- Crossover group 2 (Experimental): Placebo first then vitamin E
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Vitamin E — Vitamin E 800IU bid

SUMMARY:
Muscular cramps are a common and uncomfortable symptom of amyotrophic lateral sclerosis (ALS). This clinical trial will compare the response of high dose vitamin E supplementation to placebo for treatment of muscular cramps in patients with ALS. We hypothesize that vitamin E will be more effective than placebo in treating cramps.

DETAILED DESCRIPTION:
This will be a single centre randomized placebo controlled crossover design trial. Participants will be randomized at study entry to protocol A (vitamin E first) or protocol B (placebo first). The first 2 weeks of the study will be a baseline assessment of the frequency, severity and duration of cramps. Patients will be blinded for the remainder of the duration of the study. For weeks 3-6 of the study, group A will receive vitamin E 800 IU bid and group B will receive placebo. For weeks 7-10 of the study, group A will receive placebo and group B will receive vitamin E. Participants will record cramp frequency and characteristics via a daily journal for the duration of the study, however the data analysis will focus on cramp frequency only during weeks 5-6 and 9-10. Weeks 3-4 and 7-8 will be used as time periods to allow the new drug to come to steady state and allow for washout of the previous drug. Data analysis will focus on the difference in cramp frequency in individual patients in each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> age 18 years)
* Probable or definite ALS by El Escorial Revised criteria
* At least 2 painful muscle cramps in one or more of the limbs per week.
* May have tried other medications for cramping in the past.
* If participants are currently on treatment for cramps and are continuing to have at least 2 cramps per week, they can be included in the trial. In this situation, the individual's previous cramp medication can be continued during the trial.
* Ideally, patients should not have any medication alterations during the duration of the trial.
* Willing to discontinue supplementary vitamin E and multivitamins containing > 400 IU of vitamin E during the trial.

Exclusion Criteria:

* Patients who are unable to safely consume the trial capsules. Individuals with significant dysphagia can be included into the study if they have a functioning PEG tube or GJ tube, through which the medication can be given.
* Patients who are unable to fill out the daily diary, either personally or via a proxy.
* Patients who have had medication changes within the last 4 weeks prior to the onset of the trial will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Reduction in number of muscle cramps experienced in a two week period. | 4 weeks

SECONDARY OUTCOMES:
Reduction in the duration of cramps and reduction in the severity of cramps | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Strong, MD, FRCPC, Principal Investigator — Clinical Neurological Sciences, London Health Sciences Centre; Christen L Shoesmith, MD, FRCPC, Study Director — Clinical Neurological Sciences, London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Steele DW, Adam GP, Saldanha IJ, Kanaan G, Zahradnik ML, Danilack-Fekete VA, Stuebe AM, Peahl AF, Chen KK, Balk EM. Postpartum Home Blood Pressure Monitoring: A Systematic Review. Obstet Gynecol. 2023 Aug 1;142(2):285-295. doi: 10.1097/AOG.0000000000005270. Epub 2023 Jun 13. PMID 37311173